CLINICAL TRIAL: NCT05198661
Title: Paraneoplastic Neurological Syndromes and Autoimmune Encephalitis Collection
Acronym: SNP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_1271
Record Dates: First submitted 2021-12-20; First posted 2022-01-20 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Paraneoplastic Neurological Syndromes or Autoimmune Encephalitis
Keywords: Paraneoplastic Neurological Syndromes; Autoimmune Encephalitis; biological collection
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System | interventions — Phosphoglycerate Dehydrogenase

STUDY DESIGN:
Intervention Model Description: Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paraneoplastic neurological syndrome patients and autoimmune encephalitis patient (Other): patients with diagnosis of paraneoplastic neurological syndrome or autoimmune encephalitis
  Interventions: Biological: Collection of biological sample with sera, CSF, buffy coat, PBMC, plasma.

INTERVENTIONS:
Biological: Collection of biological sample with sera, CSF, buffy coat, PBMC, plasma. — Blood is collected only one time by blood sample to obtain serum, buffy coat, plasma and PBMC.
  2 *4ml of blood on dry tube 2 *4ml of blood on EDTA tube If possibility of delivery in 48 hours at the Centre of Biological Resources, 7*4ml of blood on heparin tube If cerebrospinal fluid has been drawn for diagnosis, remaining sample available will be stored in the collection

SUMMARY:
Numerous neurological disorders affecting the central and peripheral nervous system can be attributed to the immune system through multiple effector mechanisms. However, current treatments could be drastically improved by faster and more accurate diagnosis. The sample collection will benefit to patients with rare neuroimmune syndromes such as Autoimmune Encephalitis (AE) and Paraneoplastic Neurological Syndromes (PNS) leading to a better and early diagnosis, as well as treatment improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patient with consent
* Patient with well-characterized antibodies in serum or cerebrospinal fluid or not
* Patient with neurological disorder compatible with PNS or auto-immune encephalitis

Exclusion Criteria:

* Refusal of consent
* Patient under guardianship

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2032-08-02 (Estimated); Study Completion 2032-08-02 (Estimated)

PRIMARY OUTCOMES:
Blood Samples | 10 years
  Assessment of biocollection of blood samples
Cerebrospinal fluid biocollection | 10 years
  Assessment of biocollection of Cerebrospinal fluid

SECONDARY OUTCOMES:
Scientific collaboration | 10 years
  Number of project issued from the biocollection
Scientific | 10 years
  Number of scientific papers issued from the biocollection

CONTACTS AND LOCATIONS:
Locations (59):
- France (59):
  - Neurology, Pointe à Pitre, Guadeloupe
  - Neurology, Aix-en-Provence
  - Neurologie, Amiens
  - Neurology, Angers
  - General neurology, Annecy
  - Neurology, Avignon
  - Neurologie, Bayonne
  - Neurology, Besançon
  - Neurology, Bobigny
  - Neurology, Bordeaux
  - Neurology, Brest
  - Intensive care medicine, Cannes
  - Neurologie, Chambéry
  - Neurology, Clermont-Ferrand
  - Neurologie, Colmar
  - Neurology, Créteil
  - General, Vascular and Degenerative Neurology, Dijon
  - Neurology, Épinal
  - Internal and general practitioner, Gap
  - Neurologie, Grenoble
  - Neurology, La Roche-sur-Yon
  - Neurology, Lille
  - Neurology, Limoges
  - Neurology, Lisieux
  - Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites autoimmunes, Lyon
  - Adult Neurology and Neuropsychology, Marseille
  - Neurologie, Marseille
  - Neurology, Marseille
  - Neurology, Mâcon
  - Neurology, Metz
  - Neurology, Montivilliers
  - General Neurology, Montpellier
  - General medicine, Mulhouse
  - Neurologie, Nancy
  - Neurology, Nantes
  - Neurologie, Nice
  - Neurology, Nîmes
  - Neurology, Paris
  - Neuropediatrics, Paris
  - Intensive Care Medicine, Paris
  - Onco-neurology, Paris
  - Neurology adult, Paris
  - Neurology, neuropsychology and language rehabilitation, Poitiers
  - Neurology, Reims
  - Neurology, Rennes
  - Vascular and general neurology, Rouen
  - Neurology, Saint-Brieuc
  - Neurology, Saint-Denis
  - Neurology, Saint-Etienne
  - Neurologie, Saint-Nazaire
  - Neurology, St-Malo
  - Neurologie, Strasbourg
  - Neurology, Strasbourg
  - Neurology, Suresnes
  - Neurology, Toulon
  - Neurologie, Tours
  - Neurology, Valenciennes
  - Neurology, Vannes
  - Neurology, Versailles

IPD SHARING:
Plan to Share IPD: Undecided